CLINICAL TRIAL: NCT03229551
Title: Xylitol Topical Irrigation for Treatment of Recalcitrant Chronic Sinusitis
Brief Title: Xylitol for Chronic Sinusitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ochsner Health System (Other)
Collaborators: Tulane University School of Medicine (Other)
Responsible Party: Principal Investigator, Edward Mccoul, MD, Physician, Ochsner Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017.317.B
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Chronic Rhinosinusitis; Rhinosinusitis; Sinusitis; Drain Sinus; Endoscopic Sinus Surgery; Biofilms; Bacterial Overgrowth
Keywords: chronic rhinosinusitis; chronically draining sinus; condemned sinus; post-endoscopic sinus surgery
MeSH Terms: conditions — Rhinosinusitis; Sinusitis | interventions — Xylitol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xylitol (Experimental): This arm will evaluate the effect of topical xylitol therapy on biofilm production with the use of PCR bacterial sequencing before and after medical intervention.
  Interventions: Drug: Xylitol
- Control (Active Comparator): This arm is the standard of care saline irrigation solution.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Xylitol — Topical 5% Xylitol (wt/vol) diluted in saline nasal irrigant. Topical corticosteroid and antibiotic as directed by bacterial DNA sequencing results will be diluted in this irrigant and administered concurrently.
  Arms: Xylitol
Drug: Saline — Saline as a standard-of-care nasal irrigant. Topical corticosteroid and antibiotic as directed by bacterial DNA sequencing results will be diluted in this irrigant and administered concurrently.
  Arms: Control

SUMMARY:
The purpose of this investigation is to conduct a randomized controlled trial within a subgroup of difficult-to-treat patients with CRS, evaluating the use of topical xylitol treatment concurrently with topical steroid/antibiotics combination in the effort to disrupt biofilms and improve disease control. The effectiveness of topical surfactants is a research gap in treating CRS but has promising correlates in other medical fields. Specifically, the investigators will be studying the effect of topical xylitol therapy on biofilm production with the use of PCR bacterial sequencing before and after medical intervention.

DETAILED DESCRIPTION:
Problem Statement:

The purpose of this investigation is to conduct a trial within a subgroup of difficult-to-treat patients with CRS. This difficult group of patients will have undergone an exhaustive surgical and medical treatment of CRS These patient often will be frustrated with the lack of improvement in their symptoms despite maximal medical and surgical therapy. The effectiveness of topical surfactants is a research gap in treating CRS but has promising correlates in other medical fields.

Purpose of Study/Potential Impact:

The purpose of this investigation is to conduct a randomized controlled trial within a subgroup of difficult-to-treat patients with CRS, evaluating the use of topical xylitol treatment concurrently with topical steroid/antibiotics combination in the effort to disrupt biofilms and improve disease control. The effectiveness of topical surfactants is a research gap in treating CRS but has promising correlates in other medical fields.

Potential Benefits:

Topical xylitol could potentially decrease CRS symptoms, leading to improvements in patient quality of life. This decrease could potentially lead to fewer visits to primary care physicians/otolaryngologists. These could lead to less antibiotics, radiographs being obtained and unnecessary surgical procedures being performed, all of which could potentially reduce the burden of medical expenditure in the treatment of this disease.

Potential Risks:

Potential risks are minimal but include a sweet aftertaste in the mouth and burning in the nose; which have been reported in previous studies.

Hypothesis:

5% (wt/vol) Xylitol saline irrigation into the diseased paranasal sinus, as a part of a post-ESS refractory CRS management plan, will reduce biofilm formation in the sinus and result in symptomatic relief in affected patients.

General Design:

A prospective, randomized, double-blinded experimental design will be utilized. Patients will be randomized into the xylitol-saline treatment arm versus the control saline arm. Concurrent corticosteroid/antibiotic therapy will be utilized in both arms based on results of bacterial DNA sequencing. Patients will undergo weekly in-office irrigations for three weeks and will be evaluated one month and three months post-treatment. The postoperative care will be standardized across all participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients above the age of 18
* History of chronic rhinosinusitis history who had undergone bilateral endoscopic sinus surgery to include at a minimum maxillary antrostomy and anterior ethmoidectomy.
* Continued chronic sinusitis that is refractory to medical therapy after surgical intervention

Exclusion Criteria:

* Patients under age of 18
* Non-English speaking
* History of immunodeficiency disease
* Cystic fibrosis
* Primary ciliary dyskinesia
* History of granulomatous disease
* Active smoker
* Treatment with antifungal medications
* Use of antifungal medications
* Acute bacterial infection requiring antibiotics
* Active pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
The effect of topical xylitol therapy on biofilm production with the use of PCR bacterial sequencing before and after medical intervention. | 3 months
  Bacterial DNA sequencing obtained via endoscopic swab will be performed pre-treatment to analyse the presence of biofims in the diseased sinus. This assay will be repeated from the same sinus post-treatment with 5% Xylitol (wt/vol) to evaluate if medical intervention decreases biofilm production in the diseased sinus.

SECONDARY OUTCOMES:
Sino-Nasal Outcome Test-22 (SNOT-22) | 3 months
  Maximum score of 110 points based on responses to 22 questions
Brief Smell Identification Test (BSIT) | 3 months
  Total scores range from 0 to 12; higher scores indicate greater olfactory function
Endoscopic appearance of the patient's sinuses in response to the use of topical xylitol | 3 months
Correlation of DNA seqeuncing results with conventional sinonasal cultures | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Data will be presented in either a paper or electronic format. Upon its arrival, it will immediately be de-identified. If presented in a paper format, it will immediately be transferred into an electronic database. Only key personnel will have access to this data. The data will be encrypted and stored on permanent hardware or within the Ochsner secure network on a password-protected workstation.

REFERENCES:
- [Background] Harvey RJ, Psaltis A, Schlosser RJ, Witterick IJ. Current concepts in topical therapy for chronic sinonasal disease. J Otolaryngol Head Neck Surg. 2010 Jun;39(3):217-31. PMID 20470665
- [Background] Al-Mutairi D, Kilty SJ. Bacterial biofilms and the pathophysiology of chronic rhinosinusitis. Curr Opin Allergy Clin Immunol. 2011 Feb;11(1):18-23. doi: 10.1097/ACI.0b013e3283423376. PMID 21150431
- [Background] Hoggard M, Wagner Mackenzie B, Jain R, Taylor MW, Biswas K, Douglas RG. Chronic Rhinosinusitis and the Evolving Understanding of Microbial Ecology in Chronic Inflammatory Mucosal Disease. Clin Microbiol Rev. 2017 Jan;30(1):321-348. doi: 10.1128/CMR.00060-16. PMID 27903594
- [Background] Rosen PL, Palmer JN, O'Malley BW Jr, Cohen NA. Surfactants in the management of rhinopathologies. Am J Rhinol Allergy. 2013 May-Jun;27(3):177-80. doi: 10.2500/ajra.2013.27.3873. PMID 23710951
- [Background] Riley P, Moore D, Ahmed F, Sharif MO, Worthington HV. Xylitol-containing products for preventing dental caries in children and adults. Cochrane Database Syst Rev. 2015 Mar 26;2015(3):CD010743. doi: 10.1002/14651858.CD010743.pub2. PMID 25809586
- [Background] Sakallioglu O, Guvenc IA, Cingi C. Xylitol and its usage in ENT practice. J Laryngol Otol. 2014 Jul;128(7):580-5. doi: 10.1017/S0022215114001340. Epub 2014 Jul 7. PMID 24999540
- [Result] Shashy RG, Moore EJ, Weaver A. Prevalence of the chronic sinusitis diagnosis in Olmsted County, Minnesota. Arch Otolaryngol Head Neck Surg. 2004 Mar;130(3):320-3. doi: 10.1001/archotol.130.3.320. PMID 15023840
- [Result] Cryer J, Schipor I, Perloff JR, Palmer JN. Evidence of bacterial biofilms in human chronic sinusitis. ORL J Otorhinolaryngol Relat Spec. 2004;66(3):155-8. doi: 10.1159/000079994. PMID 15316237
- [Result] Antunes MB, Feldman MD, Cohen NA, Chiu AG. Dose-dependent effects of topical tobramycin in an animal model of Pseudomonas sinusitis. Am J Rhinol. 2007 Jul-Aug;21(4):423-7. doi: 10.2500/ajr.2007.21.3046. PMID 17882910
- [Result] Chiu AG, Antunes MB, Palmer JN, Cohen NA. Evaluation of the in vivo efficacy of topical tobramycin against Pseudomonas sinonasal biofilms. J Antimicrob Chemother. 2007 Jun;59(6):1130-4. doi: 10.1093/jac/dkm087. Epub 2007 Apr 3. PMID 17405780
- [Result] Brown CL, Graham SM, Cable BB, Ozer EA, Taft PJ, Zabner J. Xylitol enhances bacterial killing in the rabbit maxillary sinus. Laryngoscope. 2004 Nov;114(11):2021-4. doi: 10.1097/01.mlg.0000147939.90249.47. PMID 15510034
- [Result] Cain RB, Lal D. Update on the management of chronic rhinosinusitis. Infect Drug Resist. 2013;6:1-14. doi: 10.2147/IDR.S26134. Epub 2013 Jan 23. PMID 23378777
- [Result] Lin L, Tang X, Wei J, Dai F, Sun G. Xylitol nasal irrigation in the treatment of chronic rhinosinusitis. Am J Otolaryngol. 2017 Jul-Aug;38(4):383-389. doi: 10.1016/j.amjoto.2017.03.006. Epub 2017 Apr 4. PMID 28390807
- [Result] Weissman JD, Fernandez F, Hwang PH. Xylitol nasal irrigation in the management of chronic rhinosinusitis: a pilot study. Laryngoscope. 2011 Nov;121(11):2468-72. doi: 10.1002/lary.22176. Epub 2011 Oct 12. PMID 21994147
- [Result] Isogangas P, Makinen KK, Tiekso J, Alanen P. Long-term effect of xylitol chewing gum in the prevention of dental caries: a follow-up 5 years after termination of a prevention program. Caries Res. 1993;27(6):495-8. doi: 10.1159/000261587. PMID 8281565
- [Result] Uhari M, Kontiokari T, Niemela M. A novel use of xylitol sugar in preventing acute otitis media. Pediatrics. 1998 Oct;102(4 Pt 1):879-84. doi: 10.1542/peds.102.4.879. PMID 9755259
- [Result] Jain R, Lee T, Hardcastle T, Biswas K, Radcliff F, Douglas R. The in vitro effect of xylitol on chronic rhinosinusitis biofilms. Rhinology. 2016 Dec 1;54(4):323-328. doi: 10.4193/Rhino15.380. PMID 27394715
- [Result] Piromchai P, Kasemsiri P, Laohasiriwong S, Thanaviratananich S. Chronic rhinosinusitis and emerging treatment options. Int J Gen Med. 2013 Jun 7;6:453-64. doi: 10.2147/IJGM.S29977. Print 2013. PMID 23785241